CLINICAL TRIAL: NCT06758635
Title: Online Versions of Single Sessions Virtual Reality (VR) Therapy and EMDR Flash Therapy on the Treatment of Flying Fear
Brief Title: Online Versions of Single Session Virtual Reality (VR) Therapy and EMDR Flash Therapy on the Treatment of Flying Fear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Haldun University (Other)
Responsible Party: Principal Investigator, Zehra Özdil Arıkan, Specialist Psychologist, Ibn Haldun University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-71395021-020-11584
Record Dates: First submitted 2024-10-03; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Fear of Flying
Keywords: fear of flying; aviophobia; virtual reality therapy; emdr therapy
MeSH Terms: conditions — Aerophobia

STUDY DESIGN:
Intervention Model Description: Accordingly, 89 people who applied voluntarily were divided into three groups randomly: a) psychoeducation and VR exposure b) psychoeducation-only. All participants were given a set of scales consisting: Clinical Global Impression Scale; FAM (Flight Anxiety Modality Questionnaire), FAS (Flight Anxiety Situations Questionnaire), and a Visual Analogue Flight Anxiety Scale (VAFAS), to assess the level of fear of flying before and one month after the treatment.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- VRET-O Group (Experimental): the participants of this group will get 3 hours lasting online single session VR therapy
  Interventions: Behavioral: Flash-O Group; Behavioral: PYSCHOEDU-O Group
- Flash-O Group (Experimental): the participants of this group will get 3 hours lasting online single session EMDR Flash therapy
  Interventions: Behavioral: VRET-O Group; Behavioral: PYSCHOEDU-O Group
- PYSCHOEDU-O Group (Placebo Comparator): the participants of this group will get 1 hour lasting online psychotherapy
  Interventions: Behavioral: VRET-O Group; Behavioral: Flash-O Group

INTERVENTIONS:
Behavioral: VRET-O Group — Arm Description: the participants of this group will get 3 hours lasting online single session VR therapy
  Other Names: single session online VRET
  Arms: Flash-O Group; PYSCHOEDU-O Group
Behavioral: Flash-O Group — Arm Description: the participants of this group will get 3 hours lasting online single session EMDR Flash therapy
  Arms: PYSCHOEDU-O Group; VRET-O Group
Behavioral: PYSCHOEDU-O Group — Arm Description: the participants of this group will get 1 hour lasting online psychotherapy
  Other Names: only psychoeducation
  Arms: Flash-O Group; VRET-O Group

SUMMARY:
The purpose of this experimental study is to explore effectiveness of Cognitive Behavioural Therapy based Virtual Reality Therapy and Eye Movement Desensitization and Reprocessing Therapy based Flash Technique compared to psychoeducation only group through developing one session online protocols. Follow up will be performed one month after the intervention.

Accordingly, 89 people who applied voluntarily were divided into three groups randomly:

1. psychoeducation and Virtual reality therapy
2. Flash technique
3. psychoeducation-only.

All participants were given a set of scales consisting:

1. The Clinical Global Impressions Scale
2. FAM (Flight Anxiety Modality Questionnaire),
3. FAS (Flight Anxiety Situations Questionnaire), and
4. Visual Analogue Flight Anxiety Scale (VAFAS), to assess the level of fear of flying before and one month after the treatment.

This work was supported by the Research Fund of Ibn Haldun University. Project Name: Online Single Session Virtual Reality Therapy Programme for Fear of Flying. Project Number: 2238.

DETAILED DESCRIPTION:
There are several therapy methods that can help individuals to overcome their flying phobia. Although traditional fear of flying exposure approaches is extensively employed, they have substantial limitations. Classical in vivo exposure for flying is not common because it is very expensive and very hard to adapt for every flight condition. Whereas VRET can give uniquely tailored exposure scenarios like air turbulence or weather conditions, in vivo exposure is harder to deliver since the therapist has little control over the scenario (Rothbaum et al., 2006). In the therapy of specific phobias, virtual reality therapy has been the most widely employed and has garnered the most empirical attention (Price et al., 2008).

While cognitive behavioral therapy (CBT) is the mainstream in the flight phobia treatment, empirical research on different psychotherapy strategies is similarly useful in the treatment of flight phobia (Triscari et al., 2015). Specific phobia studies on the Eye Movement Desensitization and Reprocessing (EMDR) therapy indicated that EMDR therapy can provide important developments within a restricted variety of sessions (De Jongh et al., 1999). The Flash technique is a new individual or group intervention technique of EMDR that aims to reduce distress and suffering related to traumatic memories quickly (Wong, 2019).

The purpose of this experimental study is to explore the effectiveness of Cognitive Behavioural Therapy based Virtual Reality Therapy and Eye Movement Desensitization and Reprocessing Therapy based Flash Technique compared to Psychoeducation only groups through developing one-session protocols.

Hypothesis

1. Is VRET-O more effective than the psychoeducation-only group for reducing participants' anxiety and avoidance behavior for fear of flying?
2. Is FLASH-O more effective than the psychoeducation-only group for reducing participants' anxiety and avoidance behaviour for fear of flying?
3. Is there any significantly meaningful decrease in post-test scores of participants' anxiety and avoidance behaviour for fear of flying when compared to the pretest scores?

Participants were blinded to which group they would be in when they started the study via the Google form link. Randomization was performed by two independent investigators according to the order of application. Randomization was performed according to the order of the list in which the participants signed the consent form. Participants were randomly assigned to one of the three groups according to the computer-generated number sequence in a 1:1:1 ratio from https://www.randomizer.org/. both study investigators and participants were blinded to the group to which they were assigned. After randomization, each participant was informed in detail about the treatment and waiting process.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65
* clinical diagnosis of fear of flying

Exclusion Criteria:

risk of suicide or self-harm,

* psychosis,
* pregnancy
* PTSD,
* recent changes for psychotropic medicine use,
* current receipt of therapy about flying phobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
FAS Test | From enrollment to the end of the follow up at 4 weeks
  The Flight Anxiety Situation Questionnaire (FAS)
VAFAS | From enrollment to the end of the follow up at 4 weeks
  A Visual Analogue Flight Anxiety Scale
FAM Test | From enrollment to the end of the follow up at 4 weeks
  The Flight Anxiety Modality Questionnaire (FAM)
Actual flight | From enrollment to the end of the follow up at 4 weeks
  Have an actual flight within 4 weeks after the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Zehra Ozdil Arikan, Istanbul, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yasar AB, Konuk E, Kavakci O, Uygun E, Gundogmus I, Taygar AS, Uludag E. A Randomized-Controlled Trial of EMDR Flash Technique on Traumatic Symptoms, Depression, Anxiety, Stress, and Life of Quality With Individuals Who Have Experienced a Traffic Accident. Front Psychol. 2022 Mar 24;13:845481. doi: 10.3389/fpsyg.2022.845481. eCollection 2022. PMID 35401305
- [Background] Van Gerwen LJ, Diekstra RF, Arondeus JM, Wolfger R. Fear of flying treatment programs for passengers: an international update. Travel Med Infect Dis. 2004 Feb;2(1):27-35. doi: 10.1016/j.tmaid.2004.01.002. PMID 17291954
- [Background] Rothbaum BO, Anderson P, Zimand E, Hodges L, Lang D, Wilson J. Virtual reality exposure therapy and standard (in vivo) exposure therapy in the treatment of fear of flying. Behav Ther. 2006 Mar;37(1):80-90. doi: 10.1016/j.beth.2005.04.004. Epub 2006 Feb 24. PMID 16942963
- [Background] Muhlberger A, Herrmann MJ, Wiedemann GC, Ellgring H, Pauli P. Repeated exposure of flight phobics to flights in virtual reality. Behav Res Ther. 2001 Sep;39(9):1033-50. doi: 10.1016/s0005-7967(00)00076-0. PMID 11520010
- [Background] Manfield PE, Taylor G, Dornbush E, Engel L, Greenwald R. Preliminary evidence for the acceptability, safety, and efficacy of the flash technique. Front Psychiatry. 2024 Jan 8;14:1273704. doi: 10.3389/fpsyt.2023.1273704. eCollection 2023. PMID 38260782
- [Background] Maltby N, Kirsch I, Mayers M, Allen GJ. Virtual reality exposure therapy for the treatment of fear of flying: a controlled investigation. J Consult Clin Psychol. 2002 Oct;70(5):1112-8. doi: 10.1037//0022-006x.70.5.1112. PMID 12362961
- [Background] Campos D, Breton-Lopez J, Botella C, Mira A, Castilla D, Mor S, Banos R, Quero S. Efficacy of an internet-based exposure treatment for flying phobia (NO-FEAR Airlines) with and without therapist guidance: a randomized controlled trial. BMC Psychiatry. 2019 Mar 6;19(1):86. doi: 10.1186/s12888-019-2060-4. PMID 30841930